CLINICAL TRIAL: NCT06347718
Title: CAR-T Cells in Systemic B Cell Mediated Autoimmune Disease
Acronym: CASTLE
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Miltenyi Biomedicine GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASTLE; 2022-001366-35 (EudraCT Number); DRKS00032279 (Registry Identifier: Deutsches Register Klinischer Studien (DRKS))
Record Dates: First submitted 2023-12-15; First posted 2024-04-04 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Systemic Lupus Erythematosus; Systemic Sclerosis; Dermatomyositis; Polymyositis
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Scleroderma, Systemic; Dermatomyositis; Polymyositis

STUDY DESIGN:
Intervention Model Description: Phase 1:
  Evaluating the safety of CAR-T-Cells in systemic autoimmune diseases with 8 patients
  Phase 2:
  Evaluating the efficiency of CAR-T-Cells in systemic autoimmune diseases with 16 patients
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Active dose (Other): A prospective, open-label, non-randomized, single-dose interventional basket study.
  Single intravenous infusion of a freshly prepared advanced therapy medicinal product (ATMP) from autologous and expanded T cells transduced ex vivo with a CD19-CAR construct.
  No control intervention (e.g. another immunosuppressive therapy). Concomitant measures: Leukapheresis and lymphodepleting therapy for conditioning.
  Interventions: Drug: anti-CD19 CAR T cell therapy

INTERVENTIONS:
Drug: anti-CD19 CAR T cell therapy — Single-dose

SUMMARY:
The investigational product is designed to effectively combat B cells in patients with autoimmune diseases. Autologous T cells enriched with CD4/CD8 are genetically engineered using a lentiviral vector to express chimeric antigen receptors (CARs) that target the CD19 antigen on the cell surface of B cells and their precursors. During treatment, patients undergo leukapheresis, lymophodepleting chemotherapy and administration of the expanded CD19-CAR-transduced T cells.

ELIGIBILITY:
Inclusion Criteria:

* General:

  * Subjects must understand and voluntarily sign an informed consent form including written consent for data protection,
  * Adults aged ≥ 18 years at time of consent,
  * Adequate renal (eGFR > 30 ml/min/m2), liver (no Child Pugh C), heart (at worst NYHA III, EF > 30%) and pulmonary (FV and DLCO > 30%) function,
  * Male subjects unless surgically sterile, must agree to use two acceptable methods for contraception (e.g. spermicide and condom) during the trial and refrain from fathering a child starting from the time of signing the Informed Consent Form (ICF) until 12 months after dosing of the IMP,
  * Females of childbearing potential (FCBP) must have a negative urine pregnancy test at screening and must agree to use a highly effective contraceptive method (Pearl in-dex <1) starting from the time of signing the ICF and for 12 months after dosing of the IMP,
  * Must be able to adhere to the study visit schedule and other protocol requirements,
  * Double vaccination against SARS-CoV-2 or SARS-CoV-2 within the last 6 months.
* SLE specific:

  * Fulfilling the 2019 ACR/EULAR classification criteria of SLE,
  * Positivity of anti-dsDNA (> 4 U/l), anti-histone (+ or more), anti-nucleosome (+ or more) or anti-Sm antibodies (+ or more),
  * Active disease at screening, defined as ≥ 1 organ system with a British Isles Lupus Assessment (BILAG) A score (severe disease activity) or ≥ 2 organ systems with a BILAG B score (moderate disease activity),
  * Insufficient response or intolerance/ contraindication to glucocorticoids and to at least 2 of the following treatments: hydroxychloroquine, mycophenolate mofetil, belimumab, methotrexate, rituximab, cyclophosphamide. Insufficient response is defined as having increased disease activity based on the definition explained in the previous bullet point.
* SSc specific:

  * Fulfilling the 2013 ACR/EULAR classification criteria of SSc),
  * Positivity (+ or more) for at least one SSc-specific parameter (Scl70, RNA polymerase, Th/To, RP11/12, U3RNP autoantibodies),
  * Signs for fast progression including (i) disease duration ≤ 5 years (from onset of first non-Raynaud manifestation), (ii) mRSS score 10-35 at screening, (iii) elevated acute phase reactant levels (CRP ≥ 6 mg/L, ESR ≥ 28mm/h or platelet count ≥ 330 G/L), (iii) mRSS increase ≥ 3 units or involvement of one new body area or mRSS increase ≥ 2 units in one body area or ≥ 1 tendon friction rub over 6 months,
  * Insufficient response or intolerance/ contraindication to at least 2 of the following treatments: mycophenolate mofetil, azathioprine, nintedanib, methotrexate, rituximab. Insufficient response is defined as having increased disease activity based on the definition explained in the previous bullet point.
* DM/PM specific:

  * Fulfilling the 2017 ACR/EULAR classification criteria for probable or definite DM or PM,
  * Presence of active myositis in muscle biopsy or muscle MRI and/or signs of interstitial lung disease related to DM/PM,
  * Positivity (+ or more) for at least one myositis-specific antibody (aminoacyl tRNA synthetases, Mi2, MDA5, SAE, SRP, ARS, HMGCR, MJ, TIF1gamma),
  * Muscle weakness as define by MMT < 142 and 2 of the following criteria: VAS patients Global ≥2cm, VAS physician Global ≥ 2cm, HAQ > 0.25, at least one muscle enzyme > 1.3 times upper limit of normal, VAS global extra muscular activity ≥ 2cm,
  * Insufficient response or intolerance/ contraindication to glucocorticoids and to at least 2 of the following treatments: mycophenolate mofetil, ciclosporin A, tacrolimus, methotrexate, rituximab, intravenous immunoglobulins. Insufficient response is defined as having increased disease activity based on the definition explained in the previous bullet point.

Exclusion Criteria:

* Clinically suitability for a less burdensome and/or approved therapeutic approach, as judged by the investigator
* ANC < 1.000/mm3, ALC < 500/mm3 or hemoglobin < 8g/dl, absolute CD3+ T cell count < 100/μl,
* Uncontrolled severe concomitant disease, such as cancer (except basal or squamous cell skin cancer) and diabetes mellitus,
* Severely impaired renal (eGFR ≤ 30 ml/min/m2), liver (Child Pugh C), heart (NYHA IV, EF ≤ 30%) and pulmonary (FV and DLCO ≤ 30%) function,
* Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if the subject were to participate in the study or confounds the ability to interpret data from the study,
* Prior treatment with anti-CD19 antibody therapy, adoptive T cell therapy or any prior gene therapy product (e.g. CAR T cell therapy),
* History of bone marrow/ hematopoietic stem cell or solid organ transplantation,
* Any concomitant severe active infection, e.g. HIV, hepatitis B or C, SARS-CoV 2 (COVID 19), or active tuberculosis as defined by a positive Quantiferon TB-test. If presence of latent tuberculosis is established then treatment according to local guidelines must have been initiated prior to enrollment,
* Diagnosis of severe neuropsychiatric SLE, inclusion body myositis or limited SSc,
* Pregnant or lactating females,
* Females who are intending to conceive during the study,
* Known hypersensitivity to any drug components,
* Malignancy in the last 5 years before screening,
* Requirement for immunization with live vaccine during the study period or within 14 days preceding leukapheresis,
* Subjects who are younger than 18 years or are incapable to understand the aim, importance and consequences of the study and to give legal informed consent,
* Have a history of alcohol or substance abuse within the preceding 6 months that, in the opinion of the Investigator, may increase the risks associated with study participation or study agent administration, or may interfere with interpretation of results,
* Subjects who possibly are dependent on the Sponsor, the Principal Investigator or other Investigators (e.g. family members).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-07-17 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
To assess the safety of anti-CD19 CAR T cell therapy in subjects with active B-driven autoimmune disease (SLE, SSc and DM/PM). | up to d 28
  Incidence and grading of severity (graded 0-4) of Cytokine Release Syndrome (CRS) and of CAR T cell-associated neurotoxicity (ICANS) within the first 4 weeks after ATMP administration.

SECONDARY OUTCOMES:
Clinical efficacy SSc | at week 24
  Overall Response Rate (ORR) at week 24 measured by specific disease activity composite indexes, each of them validated for the specific disease:
  SSc: No progression of interstitial lung disease with worsening of FVC1 (>10 percentage) or worsening of FVC1 (5-10 percentage) plus increase in respiratory symptoms or worsening of FVC1 (5-10 percentage) plus progression of high-resolution computed tomography changes after 24 weeks.
Clinical efficacy SLE | at week 24
  Overall Response Rate (ORR) at week 24 measured by specific disease activity composite indexes, each of them validated for the specific disease:
  SLE: Fulfillment of DORIS remission criteria of SLE at week 24.
Clinical efficacy DM | at week 24
  Overall Response Rate (ORR) at week 24 measured by specific disease activity composite indexes, each of them validated for the specific disease:
  DM: 2016 ACR/EULAR moderate or major response.
Cellular response | up to week 24
  * amount of CAR T cells in the peripheral blood (cells/µl)
  * amount of B cells in the peripheral blood (cells/µl)
  * expansion of CAR T cells in the patient over time in cells/µl
Serological response | up to week 24
  Levels of respective serum autoantibodies at week 24 including incidence of sero-conversion measured in IE/ml
  * SLE: ANA-Titer, anti-dsDNA, anti-nucleosomes, anti-Sm, anti-cardiolipin IgG, C3 (mg/dl), C4 (mg/dl)
  * SSc: ANA-Titer, anti-SCL70, anti-RNA polymerase III, anti-topoisomerase
  * DM: ANA-Titer, anti-Mi2, anti-Tif1, anti-MDA5, anti-Jo1, anti-NXP2
Success of IMP process | up to week 24
  Success of the manufacturing process by GMP certification of the product (in percentage)
Physicians Global Assessment to measure quality of life | up to week 24
  Physician's Global Assessment (PhGA) of disease activity (VAS 0-100mm), (0=no disease activity, 100=worst disease activity)
Patient's Global Assessment to measure quality of life | up to week 24
  Patient's Global Assessment (PtGA) of disease activity (VAS 0-100mm), (0=no disease activity, 100=worst disease activity)
Health Assessment Questionnaire | up to week 24
  Disease Index HAQ-DI (0-4 per question; 0=best function, 4=worst function)
Functional Assessment of Chronic Illness Therapy | up to week 24
  Fatigue with FACIT Fatigue questionaire, from 8-44, (8=worst, 44=best, serious fatigue defined <30)
SLE-specific disease activity over time per subject | up to week 24
  British Isles Lupus Assessment Group (BILAG) index Improvement of organ involvement according to BILAG A-E (A=severe organ involvement, E=mild organ involvement)
SSc-specific disease activity over time per subject | up to week 24
  modified Rodnan Skin Score (mRSS) points 0-4 according to skin stiffness (0=no thickening, 3=severe thickening)
DM/PM-specific disease activity over time per subject | up to week 24
  Physician's global assessment (PhGA) of extramuscular activity 0-100mm (0=no disease activity, 100=worst disease activity)
SLE-specific disease activity over time per subject | up to 24 weeks
  Systemic Lupus Erythematosus Disease Activity Index (SLEDAI) points 1-8 according to organ involvement 1=mild organ involvement, 8=severe organ involvement)
DM/PM-specific disease activity over time per subject | up to 24 weeks
  Manual Muscle Testing (MMT) points 0-150 (0=paraplegia, 150=full muscle strength)

CONTACTS AND LOCATIONS:
Overall Officials: Georg Schett, Prof. Dr. med. univ., Principal Investigator — Universitätsklinikum Erlangen
Locations (1):
- Universitätsklinikum Erlangen, Erlangen, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Muller F, Hagen M, Wirsching A, Kharboutli S, Aigner M, Volkl S, Kretschmann S, Tascilar K, Taubmann J, Bucci L, Raimondo MG, Bergmann C, Rothe T, Corte G, Tur C, Munoz L, Boltz S, Schuster L, Hartmann F, Garantziotis P, Sporl S, Vasova I, Gerbitz A, Spriewald B, Kiener H, Giannarelli D, Locatelli F, D'Agostino MA, Hanssens L, Miltenyi S, Bozec A, Grieshaber-Bouyer R, Mackensen A, Schett G. CD19 CAR-T cells for treatment-refractory autoimmune diseases: the phase 1/2 CASTLE basket trial. Nat Med. 2026 Jan 7. doi: 10.1038/s41591-025-04185-6. Online ahead of print. PMID 41501497